CLINICAL TRIAL: NCT04051255
Title: Influence of Smoking on Clinical, Microbiological and Immunologic Parameters in Patients With Aggressive Periodontitis Treated With Non-surgical Mechanical Therapy Associated With Systemic Antibiotic Therapy.
Brief Title: Influence of Smoking on Clinical, Microbiological and Immunologic Parameters in Patients With Aggressive Periodontitis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Renato Casarin, Professor of Periodontics in Piracicaba Dental School-FOP/UNICAMP, University of Campinas, Brazil
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 088325/2017
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Periodontal Diseases; Aggressive Periodontitis
MeSH Terms: conditions — Periodontal Diseases; Aggressive Periodontitis | interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Smokers aggressive periodontits (Experimental): The patients were treated by a single-session of periodontal debridement under local anaesthesia during 45 minutes, using an ultrasonic instrument#, using subgingival tips* and irrigation with sterile saline solution, by the same operator (MGC, Paulista University, São Paulo, Brazil). After the debridement, all patients has prescribed with Amoxicillin 500 mg and Metronidazole 400 mg, every 8 hours, for 10 days (Casarin et al., 2012). Subjects were extensively informed about the intake of the prescribed medication. Subjects were clinically and microbiologically monitored at baseline (before therapy) and at 3 and 6 months post-therapy. During the monitored sessions, oral hygiene was evaluated and home care instructions were re-emphasized. Additionally, all subjects were recalled monthly for oral hygiene instructions.
  Interventions: Drug: full mouth ultrassonic debridement associated to Amoxicilin 500 + Metronidazole 400 mg
- Non-smokers aggressive periodontits (Experimental): The patients were treated by a single-session of periodontal debridement under local anaesthesia during 45 minutes, using an ultrasonic instrument#, using subgengival tips* and irrigation with sterile saline solution, by the same operator (MGC, Paulista University, São Paulo, Brazil). After the debridement, all patients was prescribed with Amoxicillin 500 mg and Metronidazole 400 mg, every 8 hours, for 10 days (Casarin et al., 2012). Subjects were extensively informed about the intake of the prescribed medication. Subjects were clinically and microbiologically monitored at baseline (before therapy) and at 3 and 6 months post-therapy. During the monitored sessions, oral hygiene was evaluated and home care instructions were re-emphasized. Additionally, all subjects were recalled monthly for oral hygiene instructions.
  Interventions: Drug: full mouth ultrassonic debridement associated to Amoxicilin 500 + Metronidazole 400 mg

INTERVENTIONS:
Drug: full mouth ultrassonic debridement associated to Amoxicilin 500 + Metronidazole 400 mg — The patients were treated by a single-session of periodontal debridement under local anaesthesia during 45 minutes, using an ultrasonic instrument#, using subgengival tips* and irrigation with sterile saline solution, by the same operator (MGC, Paulista University, São Paulo, Brazil). After the debridement, all patients was prescribed with Amoxicillin 500 mg and Metronidazole 400 mg, every 8 hours, for 10 days (Casarin et al., 2012). Subjects were extensively informed about the intake of the prescribed medication. Subjects were clinically and microbiologically monitored at baseline (before therapy) and at 3 and 6 months post-therapy. During the monitored sessions, oral hygiene was evaluated and home care instructions were re-emphasized. Additionally, all subjects were recalled monthly for oral hygiene instructions.

SUMMARY:
Treatment of smoker patients with AgP is considered a challenge to periodontists. To date, only one controlled clinical study (De Genaro Modanese et al., 2016) evaluated the effect of full mouth ultrasonic debridment (FMUD) on smokers with aggressive periodontitis. Its results showed significant improvements in clinical parameters (plaque index PI, bleeding on probing- BoP and probing depth-PD), and immunologic (reductions in interleukin 6- IL-6, tumor necrosis factor- α TNF-α levels), although the results were more favorable for non-smoking patients. Antimicrobials associated to mechanical therapy has been extensively studied (Hafajee et al., 2003, Heitz-Mayfield, 2006). The association of Amoxicillin and Metronidazole have had good clinical and microbiological results in randomized clinical trials in the treatment of AgP (Casarin et al., 2012, Sgolastra et al., 2012, Keestra et al., 2015).

Thus, this study investigates clinical, microbiological and immunological influence of smoking in the periodontal debridement associated to Amoxiciclin and Metronidazole of young individuals with pronounced periodontal destruction, compared with non-smokers individuals.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of generalized aggressive periodontitis, according to the American Academy of Periodontology-AAP, 1999;
* presence of at least 15 teeth;
* presence of at least 6 teeth containing 6 deep sites (≥ 7 mm), which are not located in bifurcation areas and
* present less than 20% of plaque index (PI) and bleeding on probing (BoP).

Exclusion Criteria:

* presence of periapical or pulpar alteration;
* presence of systemic alteration or use of medications (6 months prior to the study) that may influence the response to periodontal treatment;
* pregnant and lactating women;
* performing periodontal treatment including subgingival instrumentation in the 6 weeks preceding the study;
* teeth with bifurcation involvement;
* teeth with marked mobility;
* oral pathology;
* history of allergy to any component of the study, and
* previous periodontal surgery in the region of interest.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level (CAL) changes at 6 months | 6 months
  Indicates the distance between the base of the gingival pocket and the cemento-enamel junction, detected with a periodontal probe of 15 mm.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campinas, UNICAMP, Piracicaba, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No